CLINICAL TRIAL: NCT04766034
Title: Impact of Behavioral Economic Strategies on Low-Income Older Adults' Food Choices in Online Retail Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-01936
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Sham Comparator): The grocery shopping simulation will not include any discounts or bundles
  Interventions: Behavioral: Simulated Grocery Shopping Exercise
- Discount (Active Comparator): The grocery shopping simulation will include discount on eligible fruits and vegetables
  Interventions: Behavioral: Simulated Grocery Shopping Exercise
- Bundles (Active Comparator): The grocery shopping simulation will include healthy bundle defaults with no discount
  Interventions: Behavioral: Simulated Grocery Shopping Exercise
- Bundles and Discount (Active Comparator): The grocery shopping simulation will include healthy bundle defaults plus a discount
  Interventions: Behavioral: Simulated Grocery Shopping Exercise

INTERVENTIONS:
Behavioral: Simulated Grocery Shopping Exercise — Participants will click a link and simulate a shopping experience by selecting a week's worth of Supplemental Nutrition Assistance Program (SNAP)-eligible groceries for their household in a web-based supermarket platform

SUMMARY:
The specific aims of this proposal are to 1) develop the components of a behavioral economics strategy (i.e., healthy bundle defaults) to influence diet behaviors; 2) characterize the online grocery shopping behaviors and attitudes of low-income adults nationally; and 3) examine the extent to which "healthy bundles defaults" and other behavioral economic strategies increase fruit and vegetable purchases among low-income adults in an online randomized controlled experiment.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-99 years
* ability to read and speak English
* have ever received SNAP benefits
* live with fewer than 5 people
* access to a personal computer, laptop, tablet, or mobile phone.

Exclusion Criteria:

* aged <18 years or >99 years
* lack the ability to read and speak English
* have never received SNAP benefits
* live with 5 or more people
* do not have access to a personal computer, laptop, tablet, or mobile phone

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7710 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Rummo, MPH, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).

REFERENCES:
- [Derived] Rummo PE, Roberto CA, Thorpe LE, Troxel AB, Elbel B. Effect of Financial Incentives and Default Options on Food Choices of Adults With Low Income in Online Retail Settings: A Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e232371. doi: 10.1001/jamanetworkopen.2023.2371. PMID 36897592

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: The grocery shopping simulation will not include any discounts or bundles
  Simulated Grocery Shopping Exercise: Participants will click a link and simulate a shopping experience by selecting a week's worth of SNAP-eligible groceries for their household in a web-based supermarket platform
- Discount: The grocery shopping simulation will include discount on eligible fruits and vegetables
  Simulated Grocery Shopping Exercise: Participants will click a link and simulate a shopping experience by selecting a week's worth of SNAP-eligible groceries for their household in a web-based supermarket platform
- Bundles: The grocery shopping simulation will include healthy bundle defaults with no discount
  Simulated Grocery Shopping Exercise: Participants will click a link and simulate a shopping experience by selecting a week's worth of SNAP-eligible groceries for their household in a web-based supermarket platform
- Bundles and Discount: The grocery shopping simulation will include healthy bundle defaults plus a discount
  Simulated Grocery Shopping Exercise: Participants will click a link and simulate a shopping experience by selecting a week's worth of SNAP-eligible groceries for their household in a web-based supermarket platform
- All Enrolled Participants - Aim 2 Survey Phase: For Aim 2, enrolled participants complete a survey prior to randomization. Those who complete the survey and remain eligible move onto Aim 3 - Randomization and Online Shopping.
Period: Aim 2 - Pre-Randomization Survey
Arm/Group | Control | Discount | Bundles | Bundles and Discount | All Enrolled Participants - Aim 2 Survey Phase
Started | 0 | 0 | 0 | 0 | 7710
Completed | 0 | 0 | 0 | 0 | 3838
Not Completed | 0 | 0 | 0 | 0 | 3872
Not completed — Never been enrolled in SNAP and/or live in a household with at least 4 people | 0 | 0 | 0 | 0 | 3752
Not completed — Did not finish survey | 0 | 0 | 0 | 0 | 120
Period: Aim 3 - Randomization/Online Shopping
Arm/Group | Control | Discount | Bundles | Bundles and Discount | All Enrolled Participants - Aim 2 Survey Phase
Started | 922 | 991 | 957 | 968 | 0
Completed | 649 | 682 | 727 | 686 | 0
Not Completed | 273 | 309 | 230 | 282 | 0
Not completed — Reused same IP address, and/or finished the survey in under one-third of median completion time | 67 | 86 | 75 | 84 | 0
Not completed — Did not finish the shopping task | 206 | 223 | 155 | 198 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Discount | Bundles | Bundles and Discount | Total
Number analyzed (Participants) | 649 | 682 | 727 | 686 | 2744
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (15.4) | 47.2 (16.1) | 47.0 (16.3) | 46.7 (16.1) | 46.7 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344 | 346 | 396 | 361 | 1447
  Male | 305 | 336 | 331 | 325 | 1297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 67 | 75 | 64 | 269
  Not Hispanic or Latino | 566 | 614 | 602 | 582 | 2364
  Unknown or Not Reported | 20 | 1 | 50 | 40 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 18 | 6 | 6 | 39
  Asian | 13 | 10 | 10 | 16 | 49
  Native Hawaiian or Other Pacific Islander | 2 | 516 | 2 | 4 | 524
  Black or African American | 99 | 91 | 93 | 107 | 390
  White | 490 | 18 | 562 | 506 | 1576
  More than one race | 16 | 28 | 4 | 7 | 55
  Unknown or Not Reported | 20 | 1 | 50 | 40 | 111
Region of Enrollment [Number; unit: participants]
  United States | 649 | 682 | 727 | 686 | 2744

OUTCOME MEASURES:

1. Primary Outcome: Real Dollars Spent on Fruit and Vegetables Per Basket
Description: "Fruits and vegetables" are defined as frozen, fresh, and canned fruits and vegetables without added sugars, fats, oils, or salt.
Time Frame: Day 1
Population: Not all participants analyzed purchased fruits and vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on fruits and vegetables.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 11.31 (12.82) | 15.27 (16.08) | 11.68 (11.36) | 14.47 (14.18)

2. Secondary Outcome: Real Dollars Spent on Eligible Fruits Only
Description: "Eligible Fruits" are defined as fruit items identified as discounted in the online store.
Time Frame: Day 1
Population: Not all participants analyzed purchased eligible fruits, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on eligible fruits.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 4.28 (7.14) | 6.51 (9.94) | 4.85 (6.78) | 6.12 (7.91)

3. Secondary Outcome: Real Dollars Spent on Eligible Vegetables Only
Description: "Eligible Vegetables" are defined as vegetable items identified as discounted in the online store.
Time Frame: Day 1
Population: Not all participants analyzed purchased eligible vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on eligible vegetables.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 7.03 (9.34) | 8.76 (11.04) | 6.84 (7.93) | 8.34 (9.94)

4. Secondary Outcome: Real Dollars Spent on Eligible Fresh Fruits and Vegetables
Description: "Eligible Fresh Fruits and Vegetables" are defined as fresh, not frozen or canned, fruit and vegetables items identified as discounted in the online store.
Time Frame: Day 1
Population: Not all participants analyzed purchased eligible fresh fruits and vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on eligible fresh fruits and vegetables.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 9.61 (11.83) | 12.94 (14.56) | 10.49 (10.67) | 12.48 (12.51)

5. Secondary Outcome: Real Dollars Spent on Eligible Frozen Fruits and Vegetables
Description: "Eligible Frozen Fruits and Vegetables" are defined as frozen fruit and vegetables items identified as discounted in the online store.
Time Frame: Day 1
Population: Not all participants analyzed purchased eligible frozen fruits and vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on eligible frozen fruits and vegetables.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 1.48 (4.01) | 2.07 (5.49) | 1.05 (3.23) | 1.83 (5.38)

6. Secondary Outcome: Real Dollars Spent on Eligible Canned Fruits and Vegetables
Description: "Eligible Canned Fruits and Vegetables" are defined as canned fruit and vegetables items identified as discounted in the online store.
Time Frame: Day 1
Population: Not all participants analyzed purchased eligible canned fruits and vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still purchase $0 or 0% of their total dollars on eligible canned fruits and vegetables.
Measure: Mean (Standard Deviation); unit: US Dollars ($)
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
US Dollars ($) | 0.22 (0.92) | 0.27 (1.20) | 0.13 (0.65) | 0.16 (0.75)

7. Secondary Outcome: Total Calories From Fruits and Vegetables Per Basket
Description: as for outcome 1
Time Frame: Day 1
Population: Not all participants analyzed purchased fruits and vegetables, as quantified in SECONDARY OUTCOME MEASURE RESULTS #8. However, all participants contributed data to this outcome as they could still contribute "0" calories from fruits and vegetables in their basket.
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
Kcal | 1298.1 (1595.0) | 1526.2 (1641.3) | 1496.8 (1472.8) | 1690.5 (1572.0)

8. Secondary Outcome: Number of Participants Who Purchased Fruits and/or Vegetables
Description: Participants who purchased fruits and/or vegetables during their online shopping trip.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Discount | Bundles | Bundles and Discount
Number analyzed (Participants) | 649 | 682 | 727 | 686
Participants | 550 | 612 | 714 | 678

9. Secondary Outcome: Number of Participants Who Kept Healthy Bundle Default Shopping Cart Items in Basket at Purchase
Description: "Healthy Bundle Default Shopping Cart Items" are defined as items placed automatically in participants' carts at the beginning of the shopping exercise. Assessed among participants in the Bundles (Arm 3) and Bundles + Discount (Arm 4) arms only.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bundles | Bundles and Discount
Number analyzed (Participants) | 727 | 686
Participants | 679 | 655

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 day per participant
Arm/Group | Control | Discount | Bundles | Bundles and Discount
All-Cause Mortality (participants affected / at risk) | 0/649 | 0/682 | 0/727 | 0/686
Serious Adverse Events (participants affected / at risk) | 0/649 | 0/682 | 0/727 | 0/686
Other Adverse Events (participants affected / at risk) | 0/649 | 0/682 | 0/727 | 0/686

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04766034/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04766034/ICF_001.pdf